CLINICAL TRIAL: NCT03058445
Title: Assessing Validity of M-Mode Time-to-Turbulence "T2T" Echo Use to Confirm CVC Tip Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: non
Record Dates: First submitted 2017-01-23; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Central Venous Cather Position
Keywords: Central venous catheter; MMode echocardiography
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main group (Experimental): This the only arm in the study Intervention: Echocariography and assessing T2T and CXR CVC tip to carina distance
  Interventions: Device: Echocardiography; Device: CVC

INTERVENTIONS:
Device: Echocardiography — Substernal 4 chamber view obtained, then MMode applied to RA, then 5ml of saline is injected
Device: CVC — Injection of 5 ml of saline

SUMMARY:
Using an ultrasound echocardiography , we will measure the time to turbulance "T2T" from injecting saline into the central venous catheter CVC to the appeareance of turbulance on the screen using an MMode. The T2T will be compared with Chest X Ray "CXR" measured distance from the tip of the CVC to the carina.

We are trying to evaluate if there is a significant correlation between the two measurements.

DETAILED DESCRIPTION:
1. Background:

   The central venous catheter (CVC) is a vital tool in the intensive care unit. It is used to provide medications, fluids nutrition and assess central venous pressure. Common sites of insertion are internal jugular and subclavian vein. It is obligatory to confirm correct positioning of the CVC in the superior vena cava (SVC) at or before the junction with the right atrium before use. The incorrectly positioned catheter can lead to significant complications including arrhythmias and haemothorax. The most common method used to confirm correct CVC tip positioning is the chest x-ray (CXR). Frequent use of CXR in intensive care leads to repeated exposure to radiation and has implications for use of resources and cost. There have been multiple attempts to develop new methods to replace the CXR for confirmation of CVC tip position without increasing patient risk of radiation.

   The use of ultrasound (US) has become routine practice to guide CVC insertion. It is well established that using ultrasound to assist in central venous catheter insertion reduces the incidence of complications (1). However ultrasound is currently not routinely used to confirm the correct position of the CVC tip.

   The correct position for the CVC tip is widely accepted to be at or slightly above the SVC junction with the right atrium. CXR is the gold standard tool for assessing the correct tip position and is routinely requested after CVC insertion in the upper body veins. Several research studies have used varied US approaches to detect CVC positioning after subclavian (SC) and internal jugular (IJ) CVC placement.. Some studies focused on the direct US identification of the distal CVC tip near to or within the right atrium or the aberrant placement within an IJ or SC vein (2) (3) (4). Others indirectly identified venous insertion and distal CVC tip location near the right atrium by the rapid entry of turbulent flow into the right atrium after agitated saline or rapid saline flush of the distal CVC port. Delayed and weak turbulence suggests aberrant venous placement whereas complete lack of turbulence is concerning for arterial CVC placement (1) (5-11).The previous studies used a 2D substernal view to detect the turbulence in the right atrium. The time measurement had no set On and Set Off on the machine , which makes it hard to review or record. A great advantage of M-mode echocardiography is its high temporal resolution which enables simple and accurate measurement of the time and distance of any structure movement.(14). We are using M-Mode to measure a temporal change which makes it a more accurate measurement. The trigger time and the end point , i.e turbulence, can be recorded , reviewed and audited.
2. Rationale of the study:

   In order to minimize the risk of radiation exposure and reduce resource use, we considered the use of Ultrasound to confirm the CVC tip position. We will assess the use of M-Mode in a novel way, we called Time to Turbulence (T2T), to determine the proximity of the CVC tip to the right atrium.

   This novel method has the potential to accurately detect the CVC tip position and may eliminate the requirement of CXR after CVC insertion if paired with chest ultrasound to exclude pneumothorax. This has the potential benefit for patients of reduced radiation exposure, faster confirmation of line position with reduced waiting time to start of medication, less requirement of patient movement to obtain the CXR and reduced cost and use of resources in radiology services.
3. Study outcome

   A. Primary outcome:

   - Correlation between T2T and CVC tip distance to right atrium (RA)

   B. Secondary outcome:
   * Effect of Height and Weight on the validity of T2T value
   * Effect of inotropic support on the validity of T2T value
   * Cut-off T2T range value to confirm CVC tip position in study population with sub-group analysis for cardiovascular parameters and inotropic support
4. Study Design:

   This is a prospective uncontrolled clinical trial. Patients will be recruited from South Tyneside District Hospital. The study data will be collected by the research team and analysed by the principal investigators.

   For this study we will recruit 25 patients based on the power of study calculation - as mentioned in the statistics section. All patients who have an upper body CVC inserted and CXR completed as part of their routine care will be eligible to be enrolled. All potential participants will be sent or given a patient information leaflet about the study. They will be approached by a member of the research team, and given the opportunity to discuss the study. If they are willing to proceed with the study, they will complete written consent forms, and baseline data will be collected. Data will be collated and analysed by the research team. For patients who lack capacity, consent will be discussed with a personal Consultee (usually their next of kin) and if agreed the patient will be enrolled into the study. Once the patient regains capacity, consent will be obtained from the patient. The patient will have the right to retrospectively withdraw from the study and all collated data will be removed from the study.

   Patients, who have CVC in place and CXR done to confirm position, will be scanned using M-Mode T2T. The Time and the CVC tip distance to carina - assessed by CXR - will be plotted on a curve to review correlation to each other.

   Variable 1: Deciding level of CVC tip on CXR:

   We used the carina level as marker for distance from CVL tip. (12)(13) Using the PAXIS screen measurement tool. The CXR that was done after the CVC inserted will be displayed on the screen. A horizontal line at the level of the carina is drawn. A perpendicular line from CVC tip to the horizontal line of the level of the Carina is drawn and measured. This measurement is (CXR measurement). If the CVC tip is above the Carina the measurement is in positive value, and if the CVC tip is below the carina the measurement is in negative value. The measurement will be in millimetres.

   Variable 2: T2T M-mode method:

   Using 5 MHz curvilinear probe the subcostal view of right atrium (RA) is obtained. M-Mode line is aligned in the centre of RA. While in M-Mode, when the scan line flips from far end of the screen to the beginning of the new screen, a 3ml bolus of saline is injected in the proximal port of the CVC. The scan is paused once the turbulence appears on the monitor in the RA area. The time from beginning of screen - the injection - to the appearance of turbulence is the "Time-To-Turbulence" (T2T). This will be recorded in seconds.

   We decided to use the proximal port - instead of the distal port which may seem more relevant - because, by this way we can detect the correlation despite the tip position is before , at , or beyond the right atrium. While if we used the distal tip , the T2T will be indifferent if the tip is before or after the RA.

   Data to be collected:

   A. Data collected before the study:
   * Age
   * Sex
   * Weight
   * Height
   * Site of the CVC
   * is CXR done to confirm position?

   B. Data to collect during the study:
   * (CXR measurement) CVC Tip to carina level
   * (M-mode measurement) T2T (3 measurements)
   * heart rhythm and rate
   * blood pressure
   * inotrope use and dose The data will be collected using a dedicated case report form (CRF). (See appendix 1)

   Inclusion Criteria:
   * Adult patients with CVC in the upper body veins:
   * Internal jugular vein (right /left)
   * Subclavian vein (right/left)
   * CXR completed to confirm CVC position

   Exclusion criteria:
   * Patient or personal Consultee refusal
   * CVC not in upper body vein
   * Inability to obtain subcostal view of RA
   * Inability to aspirate blood from distal lumen of CVC
5. Statistics and data analysis:

Statistician Mr. Paul Bassett will do our data analysis. We will use Linear Regression to detect whether the CXR measurement variable is associated with the T2T measurement variable. If a strong correlation is found we will find an equation that describes the relationship and can be used to predict the CXR measurement value from T2T measurement.

To detect correlation of 0.6 or above, with a 5% significance level and 90% power, would require a sample size of 25.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with CVC in the upper body veins:

  * Internal jugular vein (right /left)
  * Subclavian vein (right/left)
  * CXR completed to confirm CVC position

Exclusion Criteria:

* - Patient or personal Consultee refusal
* CVC not in upper body vein
* Inability to obtain subcostal view of RA
* Inability to aspirate blood from distal lumen of CVC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between T2T and CVC tip distance to right atrium (RA) | 6 months

SECONDARY OUTCOMES:
Correlation between T2T fractioned to the patient's height in meters and CVC tip distance to right atrium (RA) | 6 months
  Effect of height on the validity of T2T value
Correlation between T2T fractioned to the patient's weight in kilograms and CVC tip distance to right atrium (RA) | 6 months
  Effect of Weight on the validity of T2T value
Comparing the correlation between T2T and CVC tip distance to right atrium (RA) in patients on inotropes to those who are not | 6 months
  Effect of inotropic support on the validity of T2T value
Cut-off T2T range in milliseconds that can confirm CVC tip position is in accepted distance in mellimeters to the carina in study population | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- South tyneside hospital, South Shields, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No